STUDY00014689 Approval: 10/13/2020 Admin Review Due: 5/4/2021 Version Date: 10122020

## **SUMMARY EXPLANATION OF RESEARCH**

Penn State College of Medicine
Penn State Health

Title of Project: Project Talk: a cluster, randomized controlled trial to engage underserved communities across the United States in advance care planning

Principal Investigator: Lauren Jodi Van Scoy, MD

Address: 500 University Drive, Hershey, PA 17033

Telephone Numbers: Weekdays: 8:00 a.m. to 5:00 p.m., 1-844-432-TALK (8255)

You are being invited to volunteer to participate in a research study. Research studies include only people who voluntarily choose to take part. This summary explains key information about this research. You are urged to ask questions about anything that is unclear to you.

- The purpose of this study is to determine whether having a group discussion about a workbook
  called the Conversation Project Starter Kit is a more effective tool for having conversations
  about medical decision-making and end-of-life issues, than other advance care planning (ACP)
  approaches.
- This study is called a randomized-control trial. Randomization means that you are put into a
  group by chance (like flipping a coin). There is no way to predict which group you will assigned
  to. There are three conversation tools (1) the Hello Game (2) The Conversation Project Starter
  Kit, and (3) Table Topics game. Your community host was randomized to the Conversation
  Project Starter Kit We will compare the information that we gather for the three tools to
  determine the usefulness of each tool.
- Anyone who attends a Project Talk event is welcome to do the Conversation Project Starter Kit
  activity as a part of the event. For those who participate in the research, you will also complete
  questionnaires. The questionnaires ask for your experience and thoughts when it comes to
  planning for medical decision-making. A notary public will be made available two weeks after
  the event for any research participant who wants to have their advance directive notarized.
- During the event, the research assistant will randomly select two tables and audio record those participants playing the Hello game. If you are seated at one of these tables and do not wish to be recorded, please let the research assistant know.
- Two weeks after the event, a research assistant will randomly select 3 4 research participants for a phone interview to ask additional questions about your game experience.
- Six months after the event, researchers will call to conduct a phone interview. During the call, you would answer questionnaires and give us any additional feedback you might have about the Conversation Project Starter Kit. You will be also be asked to verify that you have completed an advance directive, and if so, to send us the signature page by using an encrypted link, secure fax or US postal mail. The phone interviews will be audio recorded.
- The expected time to complete these activities is:

The Conversation Starter Kit group discussion
 Research questionnaires:
 Follow-up interview at 2 weeks (if you are selected)
 15 - 20 minutes

STUDY00014689 Approval: 10/13/2020 Admin Review Due: 5/4/2021 Version Date: 10122020

Follow-up phone interview at 6 months

o Advance Directive verification

20 -30 minutes 5 minutes

- You may opt not to participate in the research and still be part of the group discussion.
- The risks that are associated with being in the research are minimal and may include distress, discomfort discussing end-of life issues, and fatigue.
- There is a risk of loss of confidentiality if your information or your identity is obtained by someone other than the investigators, but precautions will be taken to prevent this from happening. The confidentiality of your electronic data created by you or by the researchers will be maintained to the degree permitted by the technology used. Absolute confidentiality cannot be guaranteed.
- Confidentiality of records are maintained by keeping your name separate from your data each
  participant is assigned a number that is kept separate from your name and not linked to your
  information. Encrypted databases are used to store all data. Audio files are deleted from recorders
  immediately after the files are uploaded to a secure storage network.
- This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena. There are some important things that you need to know about the Certificate of Confidentiality.
  - The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.
  - Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.
- The benefits of participating in this study may include you becoming better prepared for medical decision-making. Society will benefit, as this research will provide important information about to help underserved Americans become better prepared for medical decision-making.
- We may use your research information in future studies without your additional informed consent. Before we use or share your information, we will remove any information that shows your identity.
- There are no costs to participate in this study.
- Research participants can receive up to \$65.00 in gift cards. A \$25.00 gift card for completing
  the questionnaires and the *Conversation Project Starter kit* activity on the event day. An
  additional \$25.00 gift card can be received after completing the 6-month follow-up phone
  interview.

STUDY00014689 Approval: 10/13/2020 Admin Review Due: 5/4/2021 Version Date: 10122020

• Research participants who are randomly selected for the 2-4-week phone interview will receive a \$15.00 gift card upon completing the call. Lunch and snacks will be provided on the day of the event. This study is funded by The National Institute on Minority Health and Health Disparities.

- The investigators have no financial relationships or conflicts of interest to disclose.
- This section is about your identifiable health information that will be collected for this research study as explained above.
  - We will use and disclose your information only as described in this summary and in the HMC privacy Notice.
  - If you do not want us to use your identifiable health information, you should not be in this
    research.
  - Your permission for the use and sharing of your identifiable health information will continue indefinitely.
  - You have the right to withdraw your permission for us to use or share your health information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing using the address on the front of this form.
  - The PSU Institutional Review Board, the Human Subjects Protection Office and the Research Quality Assurance Office at HMC/PSU, the sponsor (if applicable), FDA (if applicable), and Office for Human Research Protections (if applicable) in the Department of Health and Human Services may need to read your medical and research records if they need to review this study as part of their duties.
  - o In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared.

You have the right to ask any questions you may have about this research. If you have questions, complaints or concerns or believe you may have been harmed from participating in this research, you should contact Dr. Lauren Jodi Van Scoy at 717-531-6704. If you have questions regarding your rights as a research subject or concerns regarding your privacy, you may contact the research protection advocate in the HMC Human Subjects Protection Office at 717-531-5687. You may call this number to discuss any problems, concerns or questions; get information or offer input.

You do not have to participate in this research. Taking part in the research study is voluntary. Your decision to participate or to decline the research will not result in any penalty or loss of benefits to which you are entitled.

Your completion of the questionnaire and research described above implies your voluntary consent to participate in the research and to allow your information to be used and shared as described above.